CLINICAL TRIAL: NCT03794791
Title: A Comprehensive HBsAg-positive Patients Centered Screening Strategy Targeting HCV(Hepatitis C) Micro-elimination (CHARSET) in Chongqing, China Establishment of a Model Toward HCV Elimination
Brief Title: A Comprehensive HBsAg-positive Patients Centered Screening Strategy
Acronym: CHARSET
Status: Completed | Type: Observational
Sponsor: Hong Ren (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Hong Ren, Principal Investigator, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: LS2018037
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis B and Hepatitis C (Disorder)
Keywords: HBV; HCV; Co-infection
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Coinfection | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- education: Education will be used to see whether or not improve the HCV screening and diagnosis in HBsAg(+) patients. Blood test ,HCV-RNA quantification test and HCV genotyping will be employed to evaluate the prevalence of HBV-HCV co-infection. Awareness of HCV infection in HBV/HCV cohort and analysis of risk factors will also be assessed.
  Interventions: Behavioral: education
- no education: There is no education at all.Screening and diagnosis of HCV infection in HBsAg(+) patients are based on voluntary. Blood test ,HCV-RNA quantification test and HCV genotyping will still be employed to evaluate the prevalence of HBV-HCV co-infection. Awareness of HCV infection in HBV/HCV cohort and analysis of risk factors will also be assessed.
  Interventions: Behavioral: no education

INTERVENTIONS:
Behavioral: education — Education Methods including video playing of HCV Introduction (disease profile, risk factors for infection, outcomes, HBV/HCV coinfection, reinfection, etc) for 5 min, booklets of relative information distribution, physicians and nurses consulting in clinic.
  Other Names: HCV RNA quantification test/HCV genotyping
  Groups: education
Behavioral: no education — Education Methods including video playing of HCV Introduction (disease profile, risk factors for infection, outcomes, HBV/HCV coinfection, reinfection, etc) for 5 min, booklets of relative information distribution, physicians and nurses consulting in clinic.
  Other Names: HCV RNA quantification test/HCV genotyping
  Groups: no education

SUMMARY:
HBV(hepatitis B virus) /HCV(hepatitis C virus) co-infection may accelerate liver disease progression and increase the risk of HCC(Hepatocellular Carcinoma)development. It is reported HCV co-infection harmfully affects liver fibrosis in HBV patients, while decompensated cirrhosis is increased in co-infected patients compared with HBV- or HCV- mono-infected patients. One meta-analysis having pooled 39 studies performed in China reported that around 5% of HCC was associated with HCV infection alone and 6% with co-infection of HBV + HCV. However, the exact prevalence of HCV infection in HBsAg(Hepatitis B virus surface antigen)(+) cohort is actually unknown. It is estimated to be between 0.7% and 16%, a percentage that varies over a wide range among several studies from literature, mainly depending on different geographical distribution and study population. However, in regions where HBV is endemic, such as China with a HBsAg positive rate of 7.18%, the probability of co-infection increases due to a similar transmission route, especially in patients with high risk of HCV infection, like dialysis, HIV infection, organ transplantation, sex workers, drug abuser, tattoo, piercing, blood donation, history of scaling or dental filling, HCV family history and so on.

As for China, the awareness of HCV infection is much lower than HBV because the occult of HCV infection, also because governments as well as medical authorities didn't input enough resources to disease education. Up to now, the national HCV elimination in China is daunting because of barriers in HCV awareness/link to care, and lack of well-established strategies. On the contrary, HBV infection has been widely known and educated to general population. As an add-on benefit, it might be relatively easier to conduct HCV screening test among those HBsAg-positive population. HCV elimination in high-risk subgroups from the basis in HBV population can be achieved with greater possibility and such model could be further shared to health care societies.

DETAILED DESCRIPTION:
1. Objective:

Primary objective:

Evaluate value of HCV education in HCV screening and diagnosis in HBsAg(+) patients

Secondary objectives:

1. Evaluate prevalence of HCV co-infection in HBV cohort in Chongqing, China
2. Assess awareness of HCV infection in HBV/HCV cohort and analysis of risk factors

2. Research methods

A. Evaluate value of HCV education in HCV screening and diagnosis in HBsAg(+) patients About 300 patients screened for HBsAg every day in the second affiliated hospital of Chongqing Medcial University. So there will be about 200,000 patients tested for HBsAg for 2 years, among which 5% is estimated to be HBsAg (+) (n=10,000) and will be informed. All of them will be asked to follow-up in Infectious Disease Department of the hospital and be divided into two groups by 1:1 randomization. Patients in the first group will not receive any disease education, but the investigators will record how many patients propose to take anti-HCV test voluntarily after those patients know the result of HBsAg test of their own (The acceptation rate of anti-HCV test is A). The second group will receive education about HCV infection as well as HBV/HCV co-infection and then be asked whether those patients are willing to do anti-HCV test or not (The acceptation rate of anti-HCV test is B). Education Methods including video playing of HCV Introduction (disease profile, risk factors for infection, outcomes, HBV/HCV coinfection, reinfection, etc) for 5 min, booklets of relative information distribution, physicians and nurses consulting in clinic. Diagnosis rate of HCV coinfection is C and D for the two groups, respectively.The investigators anticipate B will be higher than A and D will be higher than C, which reflects impact from disease education. Considering some patients with HBsAg(+) might not be willing to be involved in the randomization part or lost to follow-up, the investigators presuppose sample size to be 3,000 for each group for evaluation importance of education.

B. Evaluate prevalence of HCV co-infection in HBV Cohort in Chongqing, China Actually all patients with HBsAg(+) (n=10,000) will be tested for anti-HCV with blood samples and the positive ones will be informed and suggested to do HCV RNA test to get an actual prevalence of HCV co-infection in HBV cohort in Chongqing.The investigators estimate about 16% of patients (1600 for 2 years) with HBsAg (+) are positive for anti-HCV, among which about 1200 patients are positive for HCV RNA test. These patients will be diagnosed as HCV infection and will go genotyping as well as link to care.

C. Awareness of HCV infection in HBV/HCV Cohort and analysis of risk factors All patients who are HBsAg(+) will be asked to finish questionnaires, including basic information, demographic information, risk factors for HBV or HCV infection (dialysis, HIV infection, organ transplantation, sex workers, drug abuser, tattoo, piercing, blood donation, history of scaling or dental filling, HCV family history and so on), awareness of their own HBV or HCV infection, etc.

3. Which, if any, policymakers will be engaged and how.

A. For Government Results of this program may enable government including public health officials to identify where to strengthen efforts. The investigators will get evidence to show the difference of screening and diagnosis rate of HCV infection between HBsAg(+) patients who received disease education and the ones who didn't. Elimination of the HCV as public health threats by 2030 might need to be based on patient education.

B. For Reimbursement Bureau So far there is not enough data on epidemiology to accurately assess potential HCV infection in HBsAg(+) patients. The entire hepatitis elimination effort depends on improving the availability of reliable data to describe the epidemiology of HCV. By executing this program the investigators will get the prevalence of HCV infection in HBsAg(+) patients in Chongqing and there is big possibility that the data is much higher than in general population.The investigators want to let the reimbursement bureau know anti-HCV and RNA test in HBsAg(+) cohort may results in better cost effectiveness in HCV diagnosis and treatment. Reimbursement in such population may be considered.

C. For Other Medical Units Two press conferences will be held at the beginning and at the end of CHARSET program to advocate the importance of increasing HCV awareness, link-to-treatment and HCV elimination. The program will also be posted on social media like WEIBO/WECHAT (something like facebook/twitter in China) and website of the second affiliated hospital of Chongqing Medical University. Because of acquisition of higher HCV screening and diagnosis rate, this model could be generalized in other medical units to benefit more patients.

4. Study Duration (in months) 24 months

ELIGIBILITY:
Inclusion Criteria:

* HBsAg(+) patients

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HBsAg(+) patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate value of HCV education | 1 Year
  This patients will receive education about HCV infection as well as HBV/HCV co-infection and then be asked whether they are willing to do anti-HCV test or not. Education Methods including video playing of HCV Introduction (disease profile, risk factors for infection, outcomes, HBV/HCV coinfection, reinfection, etc) for 5 min, booklets of relative information distribution, physicians and nurses consulting in clinic.

SECONDARY OUTCOMES:
Prevalence of HCV co-infection | 1 Year
  All patients with HBsAg(+) (n=10,000) will be tested for anti-HCV with blood samples and the positive ones will be informed and suggested to do HCV RNA test to get an actual prevalence of HCV co-infection in HBV cohort in Chongqing. The investigators estimate about 16% of patients (1600 for 2 years) with HBsAg (+) are positive for anti-HCV, among which about 1200 patients are positive for HCV RNA test. These patients will be diagnosed as HCV infection and will go genotyping as well as link to care.
Awareness of HCV infection | 1 Year
  All patients who are HBsAg(+) will be asked to finish questionnaires, including basic information, demographic information, risk factors for HBV or HCV infection (dialysis, HIV infection, organ transplantation, sex workers, drug abuser, tattoo, piercing, blood donation, history of scaling or dental filling, HCV family history and so on), awareness of their own HBV or HCV infection, etc.

CONTACTS AND LOCATIONS:
Overall Officials: HONG REN, Prof., Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The 2nd affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pol S, Haour G, Fontaine H, Dorival C, Petrov-Sanchez V, Bourliere M, Capeau J, Carrieri P, Larrey D, Larsen C, Marcellin P, Pawlostky JM, Nahon P, Zoulim F, Cacoub P, de Ledinghen V, Mathurin P, Negro F, Pageaux GP, Yazdanpanah Y, Wittkop L, Zarski JP, Carrat F; French Anrs Co22 Hepather Cohort. The negative impact of HBV/HCV coinfection on cirrhosis and its consequences. Aliment Pharmacol Ther. 2017 Dec;46(11-12):1054-1060. doi: 10.1111/apt.14352. Epub 2017 Oct 9. PMID 28994127
- [Background] Wang M, Wang Y, Feng X, Wang R, Wang Y, Zeng H, Qi J, Zhao H, Li N, Cai J, Qu C. Contribution of hepatitis B virus and hepatitis C virus to liver cancer in China north areas: Experience of the Chinese National Cancer Center. Int J Infect Dis. 2017 Dec;65:15-21. doi: 10.1016/j.ijid.2017.09.003. Epub 2017 Sep 19. PMID 28935244
- [Background] Papadopoulos N, Papavdi M, Pavlidou A, Konstantinou D, Kranidioti H, Kontos G, Koskinas J, Papatheodoridis GV, Manolakopoulos S, Deutsch M. Hepatitis B and C coinfection in a real-life setting: viral interactions and treatment issues. Ann Gastroenterol. 2018 May-Jun;31(3):365-370. doi: 10.20524/aog.2018.0255. Epub 2018 Mar 28. PMID 29720863
- [Background] Wang H, Swann R, Thomas E, Innes HA, Valerio H, Hayes PC, Allen S, Barclay ST, Wilks D, Fox R, Bhattacharyya D, Kennedy N, Morris J, Fraser A, Stanley AJ, Gunson R, Mclntyre PG, Hunt A, Hutchinson SJ, Mills PR, Dillon JF. Impact of previous hepatitis B infection on the clinical outcomes from chronic hepatitis C? A population-level analysis. J Viral Hepat. 2018 Aug;25(8):930-938. doi: 10.1111/jvh.12897. Epub 2018 Apr 15. PMID 29577515
- [Background] Lazarus JV, Wiktor S, Colombo M, Thursz M; EASL International Liver Foundation. Micro-elimination - A path to global elimination of hepatitis C. J Hepatol. 2017 Oct;67(4):665-666. doi: 10.1016/j.jhep.2017.06.033. Epub 2017 Jul 29. No abstract available. PMID 28760329
- [Derived] Cai D, Zhang D, Hu P, Ren H. A Comprehensive Hepatitis B Surface Antigen-Positive Patient-Centered Screening and Linkage to Care Strategies Targeting Microelimination of Hepatitis C Virus Infection in Chongqing, China. Can J Gastroenterol Hepatol. 2022 Dec 27;2022:9644576. doi: 10.1155/2022/9644576. eCollection 2022. PMID 36606100